CLINICAL TRIAL: NCT07251608
Title: Randomized, Open-Label, Safety Pilot Study of Multiple Subcutaneous and Intramuscular Injections of Niagen® Plus
Brief Title: Randomized, Open-label, Safety Study of Subcutaneous and Intramuscular Injections of Niagen® Plus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ChromaDex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IH-NP-101
Record Dates: First submitted 2025-11-03; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1:1:1 into four parallel arms receiving Niagen®Plus by either subcutaneous or intramuscular injection at two dose levels (50 mg or 100 mg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50 mg Subcutaneous Niagen®Plus (Experimental): Participants receive 50 mg Niagen®Plus administered subcutaneously (under the skin) once daily for three consecutive days during in-clinic visits (Days 1-3). Participants then continue self-administered subcutaneous injections of the same dose three times per week (Monday, Wednesday, Friday) from Days 10-100.
  Interventions: Drug: Niagen®Plus
- 100 mg Subcutaneous Niagen®Plus (Experimental): Participants receive 100 mg Niagen®Plus administered subcutaneously once daily for three consecutive days during in-clinic visits (Days 1-3). Participants then continue self-administered subcutaneous injections of the same dose three times per week (Monday, Wednesday, Friday) from Days 10-100.
  Interventions: Drug: Niagen®Plus
- 50 mg Intramuscular Niagen®Plus (Experimental): Participants receive 50 mg Niagen®Plus administered intramuscularly (into the deltoid muscle) once daily for three consecutive days during in-clinic visits (Days 1-3). No further at-home injections are performed; participants return for follow-up visits on Days 10, 40, and 100.
  Interventions: Drug: Niagen®Plus
- 100 mg Intramuscular Niagen®Plus (Experimental): Participants receive 100 mg Niagen®Plus administered intramuscularly (into the deltoid muscle) once daily for three consecutive days during in-clinic visits (Days 1-3). No further at-home injections are performed; participants return for follow-up visits on Days 10, 40, and 100.
  Interventions: Drug: Niagen®Plus

INTERVENTIONS:
Drug: Niagen®Plus — Pharmaceutical-grade nicotinamide riboside chloride (NRCl), compounded for sterility and reconstituted in bacteriostatic water for injection. Administered by subcutaneous or intramuscular injection at 50 mg or 100 mg per dose. Participants receive three clinician-administered injections during clinic visits on Days 1-3, followed by at-home subcutaneous self-administration three times per week (Monday, Wednesday, Friday) from Days 10-100, depending on study arm.

SUMMARY:
The goal of this study is to learn about the safety of Niagen®Plus, an injectable form of nicotinamide riboside (NR), and to see how it affects levels of NAD+ in the blood. Niagen®Plus will be given either by subcutaneous (under the skin) or intramuscular (into the muscle) injection at two dose levels (50 mg or 100 mg).

The main questions this study aims to answer are:

Is Niagen®Plus safe and well-tolerated when given by injection several times over 100 days?

How do NAD+ levels in blood change after repeated doses of Niagen®Plus?

What are participants' and clinicians' experiences with the injections?

Researchers will also look at changes in fatigue, sleep, quality of life, inflammation markers, mitochondrial efficiency, and perceived skin appearance.

Participants will:

Receive three injections in clinic on Days 1-3, followed by a Day 10 follow-up visit

Self-inject Niagen®Plus at home three times per week from Days 10-100

Return to the clinic on Days 40 and 100 for safety and laboratory testing

Complete short surveys about fatigue, sleep, and overall well-being throughout the study

The study will include 40 generally healthy adults and will last about 100 days per participant.

DETAILED DESCRIPTION:
This is a single-site, prospective, randomized, open-label, parallel 4-arm pilot trial designed to evaluate the safety and pharmacodynamic effects of Niagen®Plus (nicotinamide riboside chloride, NRCl) when administered by injection. The study includes two phases over approximately 100 days per participant.

In Phase 1, participants receive three consecutive daily injections of Niagen®Plus (50 mg or 100 mg; subcutaneous or intramuscular) administered in clinic on Days 1-3, followed by a Day 10 follow-up visit for safety evaluation and laboratory testing. In Phase 2, participants continue self-administration of subcutaneous Niagen®Plus at home three times per week (Monday, Wednesday, Friday) through Day 100, returning to the clinic on Days 40 and 100 for repeat safety assessments, sample collection, and exploratory analyses.

Primary endpoints assess safety and tolerability through vital signs, comprehensive metabolic and hematologic panels (CMP, CBC, homocysteine), and adverse-event monitoring. Secondary endpoints include changes in whole-blood NAD⁺ concentrations measured by dried-blood-spot analysis and clinician- and participant-reported injection experience. Exploratory endpoints include fatigue, energy, sleep, and quality-of-life assessments; plasma biomarkers of inflammation (C-reactive protein); phenotypic age calculation; oxidative stress testing (in urine); mitochondrial efficiency testing; and subjective evaluations of skin appearance.

The target enrollment is 40 generally healthy adults (10 per arm). The study is not powered for hypothesis testing but will inform the design of subsequent placebo-controlled trials by characterizing safety profiles, pharmacokinetic trends, and feasibility of at-home administration.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults, aged 18+
* Demonstrated baseline fatigue as determined by a below average score from the FAS (threshold prespecified in SAP).
* NAD+ or NAD+ precursor injection naïve (including intravenous, intramuscular, subcutaneous, or other injection route) (i.e., 8 weeks abstinent)
* Non-anemic
* Willingness to adhere to lifestyle considerations and study procedures.
* Ability to read English, and provide written informed consent.
* Willingness to self-administer the study material, via subcutaneous injection for 90 days (days 10-100 of the study), and complete finger prick blood collections.

Exclusion Criteria:

* One or more uncontrolled chronic illness including but not limited to diabetes, cardiovascular disease, liver, disease, kidney disease, or any form of cancer. An uncontrolled chronic illness, in this case, is defined as any changes to medication or other treatment modalities in the last 90 Days.
* More than one chronic disease diagnosis under active treatment.
* Any chronic disease, as determined by the primary investigator, that increases risk or confounds safety.
* Any acute illness within 14 Days prior to Visit 1 (Day 1).
* Cancer diagnosis within the last 5 years
* Anemia (as defined by hemoglobin levels below 100 g/L, and other blood measures)
* Current pregnancy or lactation; unwilling to use effective contraception if of childbearing potential.
* Use of any NAD+ supplement, NAD+ precursor, or vitamin B3 product, orally, nasally, by patch, or injection within the last 60 Days. NAD+ precursors and related compounds include niacin (NA), nicotinamide (NAM), nicotinamide riboside (NR), nicotinamide mononucleotide (NMN), NAD+, NADH, NAD+3, inositol hexanicotinate, apigenin; etc. The exception is the use of a daily oral multivitamin, that may contain vitamin B3 (niacin/nicotinamide). Such use will need to be documented.
* Hypersensitivity or allergy to NR, niacin, other forms of vitamin B3/NAD+ precursors, bacteriostatic water
* Significant aversion to needles or finger pricks.
* Participation in another clinical intervention study, 90 Days (or 5 half-lives of the intervention, whichever is longer) prior to Visit 1 (Day 1).
* Any other condition rendering the participant unsuitable per investigator.
* Excessive daily use of alcohol, defined as 4 or more drinks on one occasion, or illicit drug use which would prevent adherence to the protocol as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From Day 1 (first injection) through Day 100 (final visit)
  The incidence and severity of treatment-associated moderate and severe adverse events (AEs) will be assessed.
Blood Pressure | Immediately before the first intervention, and through the 100th day of the study.
  Blood pressure, systolic and diastolic, will be measured
Heart Rate | Immediately before the intervention and through the 100th day of the study (final visit).
  Heart rate will be measured.
Pulse Rate | Immediately before and through the 100th day of the study (final visit).
  Pulse rate will be measured.
Respiratory Rate | Immediately before and through the 100th day of the study (final visit).
  Respiratory rate will be measured.
Blood Oxygen | Immediately before and through the 100th day of the study (final visit).
  Blood oxygen level will be measured.
Complete Blood Count | Immediately before and through the 100th day of the study (final visit).
  A complete blood count with differential will be evaluated through whole blood samples
Comprehensive Metabolic Panel | Immediately before and through the 100th day of the study (final visit).
  Comprehensive metabolic panel will be evaluated through whole blood samples
Homocysteine | Immediately before and through the 100th day of the study (final visit).
  Homocysteine will be measured from venous blood samples as part of the primary safety laboratory panel. Levels will be analyzed as absolute values and change-from-baseline to evaluate any clinically significant elevations or shifts associated with repeat dosing of Niagen®Plus.
High-Sensitivity C-Reactive Protein (hs-CRP) | Immediately before and through the 100th day of the study (final visit).
  High-sensitivity C-reactive protein will be assessed from venous blood samples as part of the primary safety laboratory panel. hs-CRP is a sensitive biomarker of systemic inflammation and may signal acute or sub-acute inflammatory responses to repeated Niagen®Plus dosing. Levels will be analyzed as absolute values and change-from-baseline to identify any clinically meaningful elevations or trends. Data will be summarized descriptively by dose and route of administration to support safety evaluation.

SECONDARY OUTCOMES:
Change in whole-blood NAD⁺ concentrations | Baseline (Day 1) through Day 100
  Quantitative change in whole-blood NAD⁺ levels measured by dried blood spot (DBS) assay at baseline and follow-up visits to characterize pharmacodynamic response to Niagen®Plus administration.
Participant- and clinician-reported injection-site experience | Immediately post-injection through 180 minutes after dosing (Days 1-3)
  Numeric rating scale (0-10) and clinician assessments of pain, erythema, swelling, and induration to characterize tolerability of subcutaneous versus intramuscular administration.

CONTACTS AND LOCATIONS:
Locations (1):
- BTT Medical Institute Aventura North, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. De-identified aggregate data and summary results will be shared with the sponsor and may be included in publications or presented at scientific meetings.

REFERENCES:
- [Background] Conze D, Brenner C, Kruger CL. Safety and Metabolism of Long-term Administration of NIAGEN (Nicotinamide Riboside Chloride) in a Randomized, Double-Blind, Placebo-controlled Clinical Trial of Healthy Overweight Adults. Sci Rep. 2019 Jul 5;9(1):9772. doi: 10.1038/s41598-019-46120-z. PMID 31278280
- See also: Commercial listing of the same compounded product (Niagen Plus injection) that is being used as the investigational product. — https://wellsrx.com/product/niagen-plus/
- See also: Laboratory assay measuring mitochondrial efficiency from dried blood spots, used as an exploratory endpoint in the study. — https://mescreen.com/pages/example-report
- See also: The current study's previous clinical trial with unpublished results. — https://clinicaltrials.gov/study/NCT06919328